CLINICAL TRIAL: NCT01920230
Title: The Effectiveness of Mindfulness Practices in the Recovery of Burnout
Acronym: Muupu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Jyvaskyla (Other)
Collaborators: Finnish Social Insurance Institution (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21000021201
Record Dates: First submitted 2013-07-29; First posted 2013-08-09 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Burnout, Professional; Stress
Keywords: Burnout; Stress; Mindfulness; Acceptance-commitment therapy (ACT); Intervention; Effectiveness; Working conditions; Work engagement; Psychological well-being; Life situation
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-ACT-intervention (Experimental): Group meetings face-to-face and web-based program using principles of mindfulness and ACT.
  Interventions: Behavioral: Mindfulness-ACT-intervention
- Control (Experimental): Control group, no intervention.
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: Mindfulness-ACT-intervention — Half of the participants (n=109) is assigned to intervention group. The intervention is based on Mindfulness-program presented by Williams & Penman (2011) and on principles of acceptance-commitment therapy (ACT). It aims to increase mindfulness skills and psychological flexibility through different exercises that are developed for improving skills of being present, dealing with thoughts and feelings as well as support clarifying individual values and value-based actions. The basic principles are presented in weekly small group meetings. Participants are guided to deepen their experiences through exercises and information that is provided via specific web-site.
  Arms: Mindfulness-ACT-intervention
Behavioral: No intervention — Half of the participants (n=109) don't get any special treatment. However the present study explores what kind of support they have had during the program.
  Arms: Control

SUMMARY:
The aim of this study is to examine the effectiveness of intervention based on mindfulness and acceptance-commitment therapy (ACT) in the recovery from job burnout. The 8-week intervention is delivered using jointly face-to-face group meetings and web-based program. The study hypothesizes that the Muupu-program is more effective than the normal practices when promoting work well-being in Finland. The participants are recruited from Finland.

DETAILED DESCRIPTION:
Mindfulness-ACT-based interventions aren't widely used in Finnish work health care a the moment. This study examines the possibility of using this kind of intervention for reducing job burnout and stress and also promoting well-being at work. Muupu-program is standardized and can be administered in varying settings. If intervention is effective, it can have an impact on Finnish practices when treating job burnout and work-related stress.

ELIGIBILITY:
Inclusion Criteria:

* Currently working
* Daily internet connection available
* Belongs to the group of most exhausted workers in Finland (BBI cut-off is set on the top 25%)

Exclusion Criteria:

* No psychological or somatic conditions or other practical reasons that hinder the possibility to participate to the program
* Acute medicine changes
* Regular psychotherapy
* Not willing to inform employer and/or work health care of participation to the study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Bergen Burnout Indicator (BBI) | Change from baseline burnout at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.
Perceived Stress Scale (PSS) | Change from baseline stress at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.

SECONDARY OUTCOMES:
Five Facet Mindfulness Questionnaire (FFMQ) | Change from baseline mindfulness at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.
Acceptance and Action Questionnaire (AAQ-II) | Change from baseline psychological flexibility at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.
Automatic Thought Questionnaire (ATQ) | Change from baseline automatic thoughts at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.

OTHER OUTCOMES:
Utrecht Work Engagement Scale (UWES) | Change from baseline work engagement at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.
Working conditions questionnaires used in Finlad | Change from baseline working conditions at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.
Depression, Anxiety and Stress Questionnaire (DASS) | Change from baseline depression, anxiety and sress at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.
Psychological Well-being (by Ryff) | Change from baseline psychological well-being at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.
Life Situation Questionnaire (LSQ, by Pulkkinen) | Change from baseline life situation at 2, 6 and 12 months
  Study has 4 time points when the same questionnaires are administered to assess possible changes in outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Puolakanaho, PhD, Principal Investigator — University of Jyväskylä, Department of Psychology; Raimo Lappalainen, PhD, Principal Investigator — University of Jyväskylä, Department of Psychology
Locations (1):
- University of Jyväskylä, Department of Psychology, Jyväskylä, Finland

REFERENCES:
- See also: Official web-page of the study — http://muupu.jyu.fi